CLINICAL TRIAL: NCT05414201
Title: A Multicenter, Open-label, Single-arm Study to Demonstrate the Efficacy and Safety of the Human Anti-TNF Monoclonal Antibody Adalimumab in Chinese Subjects Requiring High Dose Corticosteroids for Active Non-Infectious Intermediate-, Posterior-, or Pan-uveitis
Brief Title: A Study to Assess Change in Disease Activity and Adverse Events of Adalimumab in Chinese Participants Requiring High Dose Corticosteroids for Active Non-Infectious Intermediate, Posterior, or Pan-Uveitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20-387
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Non-infectious Intermediate Posterior- or Pan-uveitis
Keywords: Humira; Adalimumab
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adalimumab (Experimental): Participants will receive a loading dose of Adalimumab 80mg SC at Baseline followed a week later by a dose of Adalimumab 40mg SC every other week.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Subcutaneous Injection
  Other Names: Humira

SUMMARY:
Non-infectious intermediate-, posterior- and pan-uveitis (NIIPPU) are sight threatening diseases with a high patient burden and negative impact on quality of life. Corticosteroids remain the mainstay of first-line treatment for NIIPPU in China despite serious side effects associated with long-term and high-dose corticosteroid use. Adalimumab is used to treat NIIPPU in adults who have had inadequate response to corticosteroids, or who need corticosteroid-sparing, or in whom corticosteroid treatment is inappropriate. The purpose of this study is to assess adverse events and effectiveness of adalimumab in Chinese participants requiring high dose corticosteroids with NIIPPU.

Adalimumab is a conditionally approved drug in China used to treat participants with NIIPPU. All participants will receive the same treatment. Approximately 87 adult participants will be enrolled at approximately 15 sites in China.

Participants will receive one subcutaneous loading dose of adalimumab at baseline followed a week later by a lower dose of adalimumab every other week for up to 30 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of Chinese descent, with full Chinese parentage.
* Diagnosed with active non-infectious intermediate uveitis, posterior uveitis, or panuveitis defined by the presence of at least 1 of the following in at least one eye:

  * Active, inflammatory chorioretinal, and/or inflammatory retinal vascular lesion
  * ≥ 2+ anterior chamber cells (Standardization of Uveitis Nomenclature [SUN] criteria); or
  * ≥ 2+ vitreous haze (National Eye Institute [NEI]/SUN criteria).
* Receiving oral prednisone from ≥ 10mg/day to ≤ 60mg/day (or oral corticosteroids equivalent) for at least two weeks before Screening and remaining on the same dose from Screening to Baseline.

Exclusion Criteria:

* Participants with the following ocular events:

  * Isolated anterior uveitis;
  * Confirmed or suspected infectious uveitis;
  * Ocular masquerade syndromes, such as ocular lymphoma;
  * Presumed ocular histoplasmosis syndrome;
  * Serpiginous choroidopathy;
  * Scleritis;
  * Corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial;
  * Macular edema as the only sign of uveitis;
  * Severe VH that precludes visualization of the fundus at the baseline visit;
  * Intraocular pressure of ≥ 25 mmHg and on ≥ 2 glaucoma medications or evidence of glaucomatous optic nerve injury;
  * Best Corrected Visual Acuity less than 20 letters Early Treatment Diabetic Retinopathy Study (ETDRS) in either eye at the Baseline visit;
  * Proliferative or severe non-proliferative diabetic retinopathy or clinically significant macular edema due to diabetic retinopathy;
  * Neovascular/wet age-related macular degeneration;
  * Abnormality of vitreo-retinal interface (i.e., vitreomacular traction, epiretinal membranes, etc.) with the potential for macular structural damage independent of the inflammatory process.
  * Ocular surgery within 90 days prior to the Baseline visit with the exception of refractive laser surgery or retinal laser photocoagulation or YAG (neodymium-doped yttrium aluminium garnet) posterior capsulotomy. These three exceptions are exclusionary within 30 days prior to Baseline.
* Previous exposure to anti-a TNF therapy inhibitor or any biologic therapy with a potential therapeutic impact on non-infectious uveitis and discontinued for reasons other than lack of efficacy or intolerance (e.g., change of insurance) is allowed after completing the specified wash-out period prior to the Baseline visit. Participants who have had lack of efficacy or intolerance to TNF inhibitors (including Humira and its biosimilars) are not eligible.
* Has received glucocorticosteroid implant, Ozurdex® (dexamethasone implant), or intravitreal adalimumab, Methotrexate (MTX) or anti-VEGF therapy at any time prior to the Baseline visit. For those with previous exposure of anti-VEGF therapy, participants must complete the specified wash-out period prior to the baseline visit.
* Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the baseline visit or oral anti-infectives within 14 days prior to the Baseline visit.
* Participant has been receiving cyclophosphamide within 30 days and initiated new cyclophosphamide treatment within 30 days prior to the Baseline visit.
* Participant treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study.
* Participant received any live vaccine with replicating potential within 28 days prior to the first dose of study drug, or expected need of live vaccination with any live vaccine with replicating potential during study participation including at least 70 days after the last dose of study drug. Live vaccines that are incapable of replicating (e.g., JYNNEOS monkeypox vaccine or Convidecia or Convidecia Air COVID-19 vaccines) are permitted.
* Participant treated with oral traditional Chinese medicine (described for the treatment of UV) within 14 day prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants that achieve quiescence in both eyes | Week 30
  Quiescence is defined as no active inflammatory chorioretinal and/or inflammatory retinal vascular lesions, anterior chamber (AC) cell grade ≤ 0.5+ and vitreous haze (VH) grade ≤ 0.5+

SECONDARY OUTCOMES:
Percentage of participants that achieve no active lesions in both eyes | Week 30
  Percentage of participants that achieve no active lesions in both eyes.
Percentage of participants that achieve Anterior Chamber (AC) cell grade ≤ 0.5+ in both eyes | Week 30
  Slit lamp examinations will be conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam will be used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria:
  Grade 0 = < 1 cell Grade 0.5+ = 1 - 5 cells Grade 1+ = 6 - 15 cells Grade 2+ = 16 - 25 cells Grade 3+ = 26 - 50 cells Grade 4+ = > 50 cells.
Percentage of participants that achieve Vitreous Haze (VH) grade ≤ 0.5+ in both eyes | Week 30
  Vitreous haze was measured using dilated indirect ophthalmoscopy (DIO) and assessed by the Investigator according to National Eye Institute (NEI) and SUN criteria:
  Grade 0: No evident vitreous haze; Grade 0.5+: Slight blurring of the optic disc margin because of the haze; normal striations and reflex of the nerve fiber layer cannot be visualized; Grade 1+: Permits a better definition of both the optic nerve head and the retinal vessels (compared to higher grades); Grade 2+: Permits better visualization of the retinal vessels (compared to higher grades); Grade 3+: Permits the observer to see the optic nerve head, but the borders are quite blurry; Grade 4+: Optic nerve head is obscured.
Percentage of participants that achieve no worsening of Best Corrected Visual Acuity (BCVA) by ≥ 15 letters on the Early Treatment Diabetic Retinopathy Study (ETDRS) in both eyes | Week 30
  Using the appropriate corrective lenses based on that visit's refraction, participant's BCVA is measured using an ETDRS chart.
Percentage of participants that achieve a ≥ 50% reduction in immunosuppression load | Week 30
  Achievement of a ≥ 50% reduction in immunosuppression load
Percentage of participants that achieve a systemic corticosteriods dose ≤ 7.5 mg | Week 30
  Achievement of a systemic corticosteriods (CS) dose of ≤ 7.5 mg

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (7):
- China (7):
  - Peking University First Hospital /ID# 243055, Beijing, Beijing Municipality
  - Shanghai General hospital /ID# 247252, Shanghai, Shanghai Municipality
  - The second affiliated hospital of Zhejiang University school of medicine /ID# 247251, Hangzhou, Zhejiang
  - Eye hospital,WMU Zhejiang Eye Hospital /ID# 247253, Wenzhou, Zhejiang
  - Beijing Tongren Hospital, CMU /ID# 243054, Beijing
  - Tianjin Medical University Eye Hospital /ID# 243056, Tianjin
  - Xi'an people's hospital/Xi'an fourth hospital /ID# 243371, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M20-387#additional-resources-section